CLINICAL TRIAL: NCT02916589
Title: The Impact of Diet on Oral Health in Overweight Individuals With Type 2 Diabetes
Brief Title: Nutrition, Oral Health and Type 2 Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kristianstad University (Other)
Responsible Party: Principal Investigator, Cecilia Widen, Researcher, Kristianstad University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2016/582
Record Dates: First submitted 2016-09-26; First posted 2016-09-27 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baseline (Placebo Comparator): The subjects will start with one week eating their normal diet.
  Interventions: Dietary Supplement: Diet
- Igelosa Diet (Active Comparator): After one week the subjects will be provided the Igelosa Diet.
  Interventions: Dietary Supplement: Diet

INTERVENTIONS:
Dietary Supplement: Diet

SUMMARY:
Obesity continues to pose major public health challenges worldwide with cardiovascular damage, hypertension and diabetes as possible subsequent conditions. The obese are at risk for mortality and morbidity as they suffer from a high level of immune sensitivity with consequences related to damage to the circulation and microvasculature. The immune process itself is modulated by cytokines, which are small proteins which can modulate the spectrum of the inflammatory process. These proteins may act as biomarkers in the mouth.

Diabetes is also a consequence of sustained obesity and this condition can strongly influence immune status. Diabetes is characterized by the failure to produce the hormone insulin or a loss of sensitivity to insulin. Without insulin high blood glucose results in the release of a series of pro-inflammatory factors, which lead to pathological processes in several organs leading to high mortality and morbidity. Periodontitis, a common complication of diabetes, is an inflammatory condition of the soft tissue of the periodontium, causing alveolar bone loss. The accessibility of the oral cavity facilitates the study of early inflammatory processes.

Changes in diet may reduce inflammation, controlling gingival inflammation as well as clinical treatment. Since 2004 Igelösa Life Science AB has developed a modified Nordic diet based on evidence, primarily from the Japanese island of Okinawa, where the world's oldest and most healthy people live. In this study we will investigate the association between Igelösa dietary intake and measurements of inflammation in 30 overweight individuals with or without other systemic diseases.

DETAILED DESCRIPTION:
Obesity and diabetes mellitus Obesity is one of our most serious public health issues (National Food Agency, 2016). In the Swedish adult (16-84 years) population, about 35% are overweight and almost 15% are obese (Statistics Sweden). The most commonly used definition of obesity is based on the body mass index (BMI; overweight 25.0-29.9 kg/m2, obesity 30.0-39.9 kg/m2 and severe obesity > 40 kg/m2) by the World Health Organization. Many studies have shown an increased risk of all-cause mortality with greater adiposity as measured by BMI. The share of overweight or obese inhabitants in Skåne has increased gradually over recent decades. Currently, more than half, (57%) of men are either overweight or obese and the corresponding figure for women is 41 percent. These obesity rates are somewhat higher than in the rest Sweden (Regional Folkhälsostrategi för Skåne, 2010). However, physical inactivity and sedentary behavior has not increased since 2000 (Regional Folkhälsostrategi för Skåne, 2010). The consequences of obesity include increased risk of coronary heart disease, high blood pressure, stroke, and diabetes.

Diabetes Diabetes is a major health problem and is characterized by elevated serum blood sugar levels (hyperglycaemia). Hyperglycemia can be the result of insulin resistance, as well as dysfunctional islet β-cells that are unable to secrete adequate insulin to regulate blood sugar levels. The financial burden to health care systems providing care to individuals with diabetes mellitus is considerable, as is the significant secondary damage to many organs of the body (Nolan et al., 2011). Recent estimates indicate that 8.3% of adults - 382 million people worldwide - have diabetes (diabetes mellitus type 1: T1D, or diabetes mellitus type 2: T2D) and this number may approach 600 million people in less than 25 years (Anonymous IDF 2013). T2D is the predominant form of the condition and accounts for at least 90% of cases. The excess global mortality in 2000 attributed to T2D, was 2.9 million deaths. In the USA, diabetes is the leading cause of blindness, as well as causing around 40% of end-stage renal failure events and 60% of non-traumatic lower-limb amputations (Nolan et al., 2011).

Periodontitis Periodontitis is a hallmark of diabetes mellitus (Loe, 1993) and is a chronic inflammatory disease of the gingiva (gum tissues), the teeth, and the supporting bone, leading to loss of connective tissue attachment to the teeth, and alveolar bone loss. The disease is a result of a complex interaction between bacteria and the host immune response (Salvi et al., 2005). Periodontal tissue destruction is caused by a host response to the development of a complex bacterial biofilm (Thomas et al., 2013). Periodontal infections trigger the release of pro-inflammatory cytokines IL1β, IL6, IL8 and TNFα, both at the site of the infection and through the endothelial cell system (Zdarilova et al., 2010; Kocgozlu et al., 2009). It is generally perceived that periodontitis is preceded by gingivitis, but the aetiology of the transition from gingivitis to periodontitis remains unknown. Gingivitis presents with swollen tissues and increased redness but with no loss of attachment of the teeth. Poor glycemic control in patients often presents with severely inflamed gum tissues and loss of tooth-supporting alveolar bone. Several studies have reported that chronic periodontitis is prevalent in patients with diabetes (Kim et al., 2013, Moodley et al., 2013). In poorly controlled type 2 diabetes pro-inflammatory cytokines and chemokines may partially explain the greater susceptibility of diabetic individuals to periodontal breakdown (Duarte et al., 2014). To identify bacterial pathogens responsible for periodontitis, one has to use both cultivation and molecular identification methods. No single or group of pathogens has been clearly identified as the causative agent or agents of gingivitis. Indeed, Kumar et al., (2003) showed 40% of organisms detected to be novel species based on ribosomal 16S cloning and sequencing. They also concluded that among the bacterial species identified in samples collected from both healthy and chronic periodontitis patients, about one third were more prevalent among non-healthy individuals. Treatment of periodontitis is usually focused on elimination of the infection by lowering the bacterial load using surgical, non-surgical or antibiotics. These treatments have considerable side effects, limited effect over time and are usually costly. However, another way to control the inflammation is through a radical change in diet.

Okinawa and Igelösa Diet Prevention of high BMI and obesity requires a range of measures including moderate dietary habits. Research show that those who consume foods rich in fiber, like whole grain, vegetables, legumes, fruit, berries and nuts, more easily retain a stable weight (National Food Agency, 2016).

Okinawa is an island in Japan that that has been top ranked in the world when it comes to longevity. The reasons behind the long lives of the original population on Okinawa is a combination of genetic and life style-related factors and it is impossible to entangle their separate roles (Steen, 2010). However, the traditional lifestyle in Okinawa is characterized by low levels of stress, natural exercise and a diet that can be described as mainly vegetarian with fish as a main source of animal protein and fat. Steen (2010) refers to the book "the Okinawa program" where the authors Suzuki, Willcox and Willcox describe "eating the Okinawa way". According to these authors food should be sourced directly from the nature, and should be made edible with as little intervention as possible. Comparable to the Swedish National Food Agency's recommendations vegetables and whole grain constitutes a large part of the natural diet, which further is characterized by its content of calcium, antioxidants in the form of flavonoids, omega-3. Another important principle is captured in the statement "weigh your options carefully" implying that most food can be consumed as long as certain foods, like animal protein and sweets are not overconsumed (Steen, 2010).

Since 2004 Igelösa Life Science AB has developed a modified Nordic diet based on evidence, primarily from the diets of the Okinawa population. The Igelösa-diet consists of food without supplements, mainly based on locally produced traditional Nordic ingredients such as intact grain (oats, rye, barley, and wheat), vegetables, legumes, root vegetables, fish, poultry, fruit and nuts. At the same time, the diet restricts the intake of sugar, red meat, delicatessen and dairy products. The diet is nutritious but contains a lower number of calories than usual recommendations.

Research within the field Changes in diet can reduce inflammation (Baumgartner et al., 2009), comparably with clinical intervention in the control of gingival inflammation (Widén et al., 2015). In 2015, a clinical nutrition study in 30 subjects with T2D was carried out in Kävlinge. For 12 weeks every individual received Igelösa diet free of charge. This consisted of two meals a day, ready to heat, including salad, fruit and snacks and breakfasts such as muesli and porridge. In the following 12 weeks individuals cooked their own food with the help of some key products. Individualized dietary advice was available. A research team at Skåne University Hospital in Malmö documented each individual's general condition and metabolic parameters of glucose, lipids and insulin. Blood, urine and faecal samples were collected at baseline and after 2, 12 and 24 weeks. The approach was effective and resulted in that several individuals no longer required insulin.

Assessment of Periodontitis Since 1963, gingival inflammation has been determined through the incidence of bleeding on probing (BOP), that is, via a slight pressure of the gums to see if it causes bleeding (Loe & Silness, 1963). BOP bias can be avoided by using state-of-the-art laser-based measurement systems which exploit the Doppler Effect to record blood flow. Laser Doppler flow readings have been shown to be positively correlated with the degree of gingival inflammation (Gleissner et al, 2006, Patiño-Marín 2005). We will apply the Doppler technique in comparison with the traditional BOP method. Cytokines (immune system signals) are biomarkers of inflammation and these can be easily measured in fluid collected from the periodontal pockets.

Aim of the Study The purpose of the study is to investigate the association between dietary intake, periodontal status, bacterial populations and measurements of inflammation in 30 obese individuals.

Specific objectives

* We wish to determine whether a change of diet leads to weight loss, a lower incidence of systemic and local inflammation, and less need for medication?
* Is this correlated with microbial population changes in the mouth?
* Is there a correlation between cytokine levels and bacterial numbers in samples of serum and gingival crevicular fluid from periodontal pockets?
* Are the Laser Doppler blood flow and measurements of pro-inflammatory cytokines better methods of assessing periodontal inflammation compared with bleeding on probing?

ELIGIBILITY:
Inclusion Criteria:

* minimum 18 teeth
* BMI>30

Exclusion Criteria:

* on anti-inflammatory medication
* current treatment with antibiotics or intake of antibiotics 3 months before participating in the study
* pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-09; Primary Completion 2016-12 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Changes in the extent of gingivitis, as determined by the severity of gingival bleeding, Before and after study procedures. | Once a week over two weeks.

SECONDARY OUTCOMES:
Change in levels of proinflammatory cytokines in serum and gingival fluid in relation to ginigival bleeding, Before and after study procedures. | Once a week over two weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Brita Larsson, Study Director — Kristianstad University
Locations (1):
- University of Kristianstad, Kristianstad, Skåne County, Sweden